CLINICAL TRIAL: NCT02088749
Title: Comparison of Weight Management Programs Delivered in Large Versus Small Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DK081607-pilot; K23DK081607 (NIH)
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Obesity
Keywords: obesity; weight loss; treatment; lifestyle
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- small group treatment (Experimental): lifestyle intervention for obesity delivered to small groups of approximately 12 participants/group
  Interventions: Behavioral: lifestyle intervention for obesity
- large group treatment (Active Comparator): lifestyle intervention for obesity delivered to a large group of approximately 30 participants
  Interventions: Behavioral: lifestyle intervention for obesity

INTERVENTIONS:
Behavioral: lifestyle intervention for obesity

SUMMARY:
The purpose of this study is to compare the 6- and 12-month weight changes associated with lifestyle interventions delivered in a large group or small groups of participants. It is hypothesized that participants receiving treatment in a small group will have greater weight loss than those assigned to a larger group.

ELIGIBILITY:
Inclusion Criteria:

* at least 21 years-old
* body mass index (BMI) between 30-45

Exclusion Criteria:

* have lost >4.5 kg in past six months
* have medical condition(s) likely to affect ability to participate in physical activity
* planning to relocate from the area in next 12 months
* unable or unwilling to attend weekly group sessions
* unwilling to accept random assignment

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change in body weight from baseline to months 6 and 12 | baseline, month 6, month 12
  Weight will be measured to the nearest 0.1 kg using calibrated digital scales at baseline, month 6, and month 12.

SECONDARY OUTCOMES:
treatment attendance | 12 months
  Participants attendance at each treatment group session was recorded.
treatment adherence | 12 months
  Participants' self-monitoring of food intake was collected to determine adherence to this component of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Dutton, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Florida State University, Tallahassee, Florida